CLINICAL TRIAL: NCT04274452
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Efgartigimod (ARGX 113) 10 mg/kg Intravenous in Adult Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study to Assess the Efficacy and Safety of Efgartigimod in Adult Patients With Primary Immune Thrombocytopenia (ITP)
Acronym: ADVANCE2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The ARGX-113-1908 study will be replaced by a similar design with a subcutaneous formulation (ARGX-113-2004)
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1908
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- efgartigimod (Experimental): Patients receiving an intravenous infusion of efgartigimod
  Interventions: Biological: efgartigimod
- placebo (Placebo Comparator): Patients receiving an intravenous infusion of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: efgartigimod — Intravenous infusion of efgartigimod
  Other Names: ARGX-113
  Arms: efgartigimod
Other: Placebo — Intravenous infusion of placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind placebo-controlled multicenter phase 3 trial to evaluate the efficacy and safety of ARGX-113 in patients with primary ITP.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the requirements of the trial and provide written informed consent (including consent for the use and disclosure of research related health information), willing and able to comply with the trial protocol procedures (including attending the required trial visits).
* Male/female aged ≥18 years at the time the informed consent form (ICF) is signed.
* Confirmed diagnosis of ITP made at least 3 months before randomization and based on the American Society of Hematology Criteria, and without a known etiology for thrombocytopenia.
* Diagnosis supported by a response to a prior ITP therapy (other than TPO RAs), in the opinion of the investigator.
* Mean platelet count of <30×10^9/L from 2 counts during the screening period including the predose count at visit 1. Additionally, a documented history of a platelet count of <30×109/L prior to screening.
* At the start of the trial, the patient either takes concurrent ITP treatment(s) and has received at least 1 prior therapy for ITP in the past, or the patient does not take treatment for ITP but has received at least 2 prior treatments for ITP. Patients receiving permitted concurrent ITP treatment(s) at baseline, must have been stable in dose and frequency for at least 4 weeks prior to randomization. Permitted concurrent ITP medications include oral corticosteroids, oral immunosuppressants, dapsone/danazol, fostamatinib, and/or oral TPO-RAs. Patients not receiving concurrent ITP therapy are also eligible for the trial if they have not received prior ITP therapy for at least 4 weeks prior to baseline, and 6 months in case of prior ITP therapy with an anti-CD20 therapy (eg, rituximab).
* Women of childbearing potential: Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before trial medication can be administered. Women must be on a stable regimen for at least 1 month of at least 1 highly effective method of contraception (ie, failure rate of less than 1% per year) during the trial and for 90 days after the last administration of the IMP.
* Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use effective contraception from signing the ICF through 90 days after the last administration of the IMP. Male patients practicing true sexual abstinence (as consistent with preferred and usual lifestyle) can be included. Sterilized male patients who have had a vasectomy and with documented absence of sperm postprocedure can be included. Male patients are not allowed to donate sperm from signing the ICF through 90 days after the last dose of the IMP.

Exclusion Criteria:

* ITP/thrombocytopenia associated with another condition, eg, lymphoma, chronic lymphocytic leukemia, viral infection, hepatitis, induced or alloimmune thrombocytopenia, or thrombocytopenia associated with myeloid dysplasia.
* Use of anticoagulants (eg, vitamin K antagonists, direct oral anticoagulants) within 4 weeks prior to randomization.
* Use of any transfusions within 4 weeks prior to randomization.
* Use of Ig (IV, subcutaneous, or intramuscular route) or plasmapheresis (PLEX), 4 weeks prior to randomization.
* Use of romiplostim within 4 weeks prior to randomization.
* Undergone splenectomy less than 4 weeks prior to randomization.
* Use of an investigational product within 3 months or 5 half-lives (whichever is longer) before the first dose of the IMP.
* Use of any monoclonal antibody within the 6 months before the first dose of the IMP.
* At the screening visit, clinically significant laboratory abnormalities as below: Hemoglobin ≤9 g/dL - OR - International normalized ratio >1.5 or activated partial thromboplastin time >1.5×ULN - OR - Total IgG <6 g/L.
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of the IMP. Patients with the following cancer can be included at any time: Adequately treated basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
* Uncontrolled hypertension, defined as a repeated elevated blood pressure exceeding 160 mmHg (systolic) and/or 100 mmHg (diastolic) despite appropriate treatments.
* History of a major thrombotic or embolic event (eg, myocardial infarction, stroke, deep venous thrombosis, or pulmonary embolism) within 12 months prior to randomization.
* History of coagulopathy or hereditary thrombocytopenia or a family history of thrombocytopenia.
* Clinical evidence of other significant serious diseases, have had a recent major surgery, or who have any other condition in the opinion of the investigator, that could confound the results of the trial or put the patient at undue risk.
* Positive serum test at screening for an active viral infection with any of the following conditions: Hepatitis B virus (HBV) that is indicative of an acute or chronic infection, Hepatitis C virus (HCV) based on HCV-antibody assay, Human immunodeficiency virus (HIV) based on test results that are associated with an acquired immunodeficiency syndrome (AIDS)-defining condition or a CD4 count <200 cells/mm3.
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases other than ITP (eg, cardiovascular, pulmonary, hematologic, gastrointestinal, endocrine, hepatic, renal, neurological, malignancy, infectious diseases, uncontrolled diabetes) despite appropriate treatments, which could put the patient at undue risk.
* Known hypersensitivity reaction to efgartigimod or 1 of its excipients.
* Previously participated in a clinical trial with efgartigimod.
* Pregnant or lactating females and those who intend to become pregnant during the trial or within 90 days after last dose of the IMP.
* Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening.
* Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of ITP or put the patient at undue risk.
* Current or history of (ie, within 12 months of screening) alcohol, drugs, or medication abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of cumulative weeks over the planned 24 week treatment period with platelet counts of ≥50×10^9/L in patients with chronic ITP. | Up to 24 weeks

SECONDARY OUTCOMES:
Number of cumulative weeks over the planned 24-week treatment period with platelet counts of ≥50×10^09/L in the overall population (chronic and persistent ITP). | Up to 24 weeks
Proportion of patients in the overall population with a sustained platelet count response defined as achieving platelet counts of ≥50×10^9/L for at least 4 of the 6 visits between week 19 and 24 of the trial | Up to 6 weeks
Proportion of patients in the overall population achieving platelet counts of ≥50×10^9/L for at least 6 of the 8 visits between week 17 and 24 of the trial | Up to 8 weeks
Proportion of patients in the overall population with overall platelet count response defined as achieving a platelet count of ≥50×10^9/L on at least 4 occasions at any time during the treatment period | Up to 24 weeks
Extent of disease control defined as the number of cumulative weeks until week 12, with platelet counts of ≥50×10^9/L in the overall population | Up to 12 weeks
Proportion of patients in the overall population with overall platelet count response defined as achieving a platelet count of ≥50×10^9/L on at least 4 occasions at any time until week 12 | Up to 12 weeks
Mean change from baseline in platelet count at each visit in the overall population. | Up to 31 weeks
Time to response defined as the time to achieve 2 consecutive platelet counts of ≥50×10^9/L in the overall population | Up to 31 weeks
The number of cumulative weeks over the treatment period with platelet counts of ≥30×10^9/L and ≥20×10^9/L above baseline in the overall population | Up to 24 weeks
In patients with baseline platelet count of <15×10^9/L, the number of cumulative weeks over the treatment period with platelet counts of ≥30×10^9/L and ≥20×10^9/L above baseline in the overall population | Up to 31 weeks
Incidence and severity of the World Health Organization (WHO)-classified bleeding events in the overall population | Up to 31 weeks
Rate of receipt of rescue therapy (rescue per patient per month) | Up to 31 weeks
Proportion of patients for whom dose and/or frequency of concurrent ITP therapies have increased at week 12 or later | Up to 24 weeks
Incidence and severity of adverse events (AEs), AEs of special interest (AESIs)and serious AEs (SAEs). | Up to 31 weeks
Vital signs, electrocardiogram (ECG), and laboratory assessments | Up to 31 weeks
Change from baseline in PRO (FACIT-Fatigue, Fact-Th6) at planned visits | Up to 31 weeks
Change from baseline in QoL (SF-36) at planned visits | Up to 31 weeks
Incidence of anti-drug antibodies (ADA) to efgartigimod | Up to 31 weeks
Pharmacokinetic parameters of efgartigimod : maximum observed serum concentration (Cmax) | Up to 31 weeks
Pharmacokinetic parameters of efgartigimod : serum concentration observed predose (Cthrough) | Up to 31 weeks
Pharmacodynamics markers: total immunoglobulin (Ig) G, IgG isotypes (IgG1, IgG2, IgG3, IgG4), antiplatelet antibody levels | Up to 31 weeks

IPD SHARING:
Plan to Share IPD: Undecided